CLINICAL TRIAL: NCT04817982
Title: Does Perineural Dexamethasone Increase the Duration of an Ulnar Nerve Block When Controlling for Systemic Effects? A Randomised, Blinded, Placebo-controlled, Paired, Non-inferiority Trial in Healthy Volunteers.
Brief Title: Does Perineural Dexamethasone Increase the Duration of an Ulnar Nerve Block When Controlling for Systemic Effects?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-138-2020
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Anesthesia, Local
Keywords: Regional anesthesia; Dexamethasone; Peripheral nerve block
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised, blinded, placebo-controlled, paired, non-inferiority trial in healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial medication will be identical in appearance and will be prepared in syringes of identical appearance with an identical volume of trial medication by an un-masked nurse who is not otherwise involved in the trial. The participant, anaesthesiologist performing the blocks, the investigators, and the outcome assessors for all outcomes will be masked to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Perineural dexamethasone (Experimental): Bilateral ulnar nerve blocks with bupivacaine. Dexamethasone will be added perineurally in this arm on the same day as the 'systemic dexamethasone' group.
  Interventions: Drug: Perineural dexamethasone
- Systemic dexamethasone (Active Comparator): Bilateral ulnar nerve blocks with bupivacaine. Placebo (saline) will be added perineurally in this arm on the same day as the 'perineural dexamethasone' group. Thereby, this ulnar nerve block will only be affected by the perineurally added dexamethasone that is absorbed and redistributed systemically.
  Interventions: Drug: Systemic dexamethasone
- Placebo (Placebo Comparator): Bilateral ulnar nerve blocks with bupivacaine. Placebo (saline) will be added perineurally in this arm on the same day as lidocaine group. This will be the actual placebo group.
  Interventions: Drug: Placebo
- Perineural lidocaine (Active Comparator): Bilateral ulnar nerve blocks with bupivacaine. Lidocaine will be added perineurally in this arm on the same day as the actual placebo group.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Perineural dexamethasone — Dexamethasone 4mg will be added perineurally to an ulnar nerve block with bupivacaine.
  Arms: Perineural dexamethasone
Drug: Lidocaine — Lidocaine 40 mg will be added perineurally to an ulnar nerve block with bupivacaine.
  Arms: Perineural lidocaine
Drug: Placebo — Saline will be added perineurally to an ulnar nerve block with bupivacaine.
  Other Names: Saline
  Arms: Placebo
Drug: Systemic dexamethasone — Dexamethasone will be added perineurally to an ulnar nerve block with bupivacaine, some will be reabsorbed and distributed systemically. Thereby, the investigators control for the systemic effects of adding perineural dexamethasone to an ulnar nerve block.
  Arms: Systemic dexamethasone

SUMMARY:
Investigators will assess if perineural dexamethasone can increase the duration of an ulnar nerve block when controlling for systemic effects in healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers will have bilateral ulnar nerve blocks performed with bupivacaine on two different days with a minimum of 14 days wash-out. On one day, the participants will also receive dexamethasone in one arm and placebo in the other. On the other day, the participants will also receive placebo in one arm and lidocaine in the other. By this using this design, the investigators will be able to assess if perineural dexamethasone can increase the duration of an ulnar nerve block when controlling for the systemic effects. Furthermore, to ensure blinding, the investigators have also incorporated the lidocaine group which also allows for the assessment of the effects of adding lidocaine to a peripheral nerve block with bupivacaine. The order of which the participant will receive dexamethasone and lidocaine will be random. It will also be random in which arm the participant receives dexamethasone and lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above
* Must fully understand the protocol and sign written informed consent
* American Society of Anaesthesiologists Physical Status Classification System of 1 or 2
* Body Mass Index above 18 kg/m^2
* For fertile women, safe contraceptives for the last month and negative urine human chorionic gonadotropin is required

Exclusion Criteria:

* Participants unable to cooperate
* Participants unable to speak or read Danish
* Age above 65 years
* Cardiovascular disease
* Allergy to study medication
* History of alcohol or substance abuse
* Intake of corticosteroids within the last 14 days
* Daily intake of prescription analgesia within the last four weeks
* Intake of over-the-counter analgesia within the last 48 hours
* Neuromuscular diseases or wounds on the arms or hands preventing adequate test or block performance.
* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Duration of the sensory nerve block, assessed by temperature discrimination (cold swab) | 24 hours
  The investigators will stimulate the skin with an alcohol swab and ask the participant if it is cold or warm. The duration of the sensory block will be defined as the time to the alcohol swab feels cold again. The investigators will assess temperature discrimination every 30 minutes.

SECONDARY OUTCOMES:
Duration of the sensory nerve block, assessed by mechanical discrimination (pinprick) | 24 hours
  The investigators will stimulate the skin with a needle. The duration of the sensory block will be defined as the time to the needle feels sharp again. The investigators will assess mechanical discrimination every 30 minutes.
Duration of analgesia, assessed by pain during tonic heat stimulation (heated thermode) | 24 hours
  The investigators will stimulate the participants' skin for 30 seconds with a thermode heated to 45 degrees Celsius. The participants rate the pain elicited on the Visual Analogue Scale using a ruler indicating "no pain" at zero millimetre on one end and "worst perceivable pain" at 100 millimetres at the opposite end. The duration of the sensory block will be defined as the time to the tonic heat stimulation elicits a painful response of Visual Analogue Scale above '0'. The investigators will assess pain every 30 minutes.
Duration of the motor block, assessed by fifth finger abduction | 24 hours
  The hand is placed facing with the volar side upwards. The hand is constricted so that only the fifth finger can abduct. The motor block is assessed using a Modified Bromage Scale. The duration of motor block is the time from block performance until Bromage grade '4' is reached or the participant indicates a feeling of normal strength in the finger.
Onset of the sensory nerve block, assessed by temperature discrimination (cold swab) | 24 hours
  The investigators will stimulate the skin with an alcohol swab and ask the participant if it is cold or warm. The onset of the sensory block will be defined as the time to the alcohol swab no longer feels cold. The investigators will assess the onset by temperature discrimination every 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Maagaard, MD, Principal Investigator — Zealand University Hospital, Køge
Locations (1):
- Zealand University Hospital, Køge, Zealand Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data will be shared upon reasonable request from researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the trial.
Access Criteria: Research project related to this trial.